CLINICAL TRIAL: NCT00167648
Title: Neoadjuvant Estradiol or Androgen Deprivation in Clinically Localized Prostate Cancer
Acronym: NE2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Pacific Northwest SPORE (Other)
Responsible Party: R. Bruce Montgomery, MD, Fred Hutchinson Cancer Research Center Pacific Northwest SPORE
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-5564-V 01
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2009-01-19 (Estimated); Status verified 2009-01

CONDITIONS: Cancer; Prostate Neoplasms
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms | interventions — Leuprolide; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Leuprolide 7.5 mg or Goserelin 3.6 mg
  Interventions: Drug: Leuprolide or goserelin
- B (Experimental): Transdermal estradiol 0.6 mg q 3 days
  Interventions: Drug: Transdermal estradiol

INTERVENTIONS:
Drug: Leuprolide or goserelin — Leuprolide 7.5 mg (4-week depot) or goserelin 3.6 mg (4-week depot)
  Arms: A
Drug: Transdermal estradiol — Estradiol patches, six at 0.1 mg each, changed every 3-4 days
  Arms: B

SUMMARY:
Prostate cancer is the most commonly diagnosed cancer among males in the U.S. More than 220,000 men will be diagnosed with prostate cancer in the USA this year and more that 31,000 will die of this disease.

Androgen deprivation, the elimination of testosterone and its active metabolites, remains the single most effective intervention available for the treatment of advanced prostate carcinoma. Androgen deprivation induces an immune response to normal prostate and prostate cancer, which is usually short-lived. Estradiol induces activation of many arms of the immune system and may be a more effective and long lasting means of inducing immunity to prostate tissue.

This study will treat clinically localized prostate cancer patients with either estrogens, or standard androgen deprivation without estrogens, prior to prostatectomy in order more completely to describe immune regulation by estradiol in men. Control tissue from patients who have not been treated with androgen deprivation will be procured from the Northwest Special Projects in Oncology Research Excellence (SPORE) tissue core and used as comparisons against the cancers treated before prostatectomy. Tumors removed at prostatectomy, tissue samples and blood samples will be assessed for immune system changes.

DETAILED DESCRIPTION:
Estrogens are effective means of treating advanced prostate cancer. In randomized studies estrogens have better cancer control rates than orchiectomy alone, suggesting that estrogen efficacy is not limited to its ability to suppress testosterone. One hypothesis is that estrogens modulate immunity to prostate cancer through direct activation of effector cells and by upregulating cytokines in prostatic stroma. Administration of estrogen in murine models induces infiltration of normal prostate with T lymphocytes even in castrate male animals potentially through induction of autoimmunity to normally cryptic prostate antigens. Estrogens activate multiple immune effectors and autoimmunity in a broad variety of experimental settings, suggesting upregulation of immune recognition on many levels. Pilot data demonstrates that estrogens upregulate expression of interferon regulated genes, major histocompatibility antigens (MHC) on prostate cancer, and increase both number and activation of natural killer (NK) cells. Other groups have shown that standard forms of androgen deprivation also induce immunity against both normal and malignant prostate tissue. We propose to test the hypothesis that administration of estrogen and/or androgen deprivation induces immune recognition of prostate cancer in humans through upregulation of major histocompatibility antigens on tumor and induction of tumor specific immunity. The specificity of estrogen effect will be tested by comparing measures of immunity in patients treated with estradiol, androgen deprivation or no neoadjuvant therapy.

Plan of therapy

The specific aims of this proposal are:

1. To treat patients with clinically localized, low to intermediate risk prostate cancer who are candidates for radical prostatectomy with either standard androgen deprivation prior to surgery (neoadjuvant androgen deprivation) or neoadjuvant transdermal estradiol. Patients will undergo radical prostatectomy 21 days after initiation of treatment.
2. To evaluate radical prostatectomy specimens obtained from these patients for expression of MHC class I and II, and NK ligands MICA and MICB in prostate carcinoma and adjacent prostate by immunohistochemistry (IHC) and Western analysis.
3. To evaluate tumor tissue for infiltration by clonal T lymphocytes, NK cells, and plasmacytoid dendritic cells using IHC and spectratyping of T cell receptor gene rearrangements.
4. To evaluate patients for the induction of tumor specific antibodies using patient immunoglobulin collected before and after neoadjuvant therapy (SEREX)
5. To evaluate patients for induction of NK cells and upregulation of the NK receptor NKG2D on patient lymphocytes by androgen deprivation and estradiol.
6. To evaluate the effects of androgen deprivation and estradiol on induction of plasma and tissue levels of interferon gamma, alpha, beta, IL-4 and GM-CSF by ELISA and ribonuclease protection assay.

ELIGIBILITY:
Inclusion Criteria:

1. Men 18 years or older with a histologic diagnosis of low to intermediate risk prostate cancer prior to radical prostatectomy as defined by:

   1. Clinical stage T1-T2b
   2. PSA < 20
   3. Gleason score < 7

   Patients who have more than one of the following prognostic factors: T2b, Gleason 7, PSA 10-20 are not eligible.
2. Patient's tumor must be considered surgically resectable as determined by a urologic evaluation
3. ECOG performance status of 0-1
4. Life expectancy greater than 2 years
5. Able to understand and give informed consent
6. Patients must agree not to take dietary phytoestrogens or other estrogen containing supplements

Exclusion Criteria:

1. Patients with locally advanced or high-risk disease as defined above.
2. Patients who have a testosterone less than 280 ng/dL.
3. Patients who have evidence of cerebrovascular accident or ischemia, recent deep venous thrombosis, pulmonary emboli, unstable angina or clinical congestive heart failure.
4. Patients who are receiving any other investigational therapy.
5. Patients with an active serious infection or other serious underlying medical condition that would otherwise impair their ability to receive protocol treatment.
6. Dementia or significantly altered mental status that would prohibit the understanding and/or giving of informed consent.
7. Patients with immunodeficiency or on oral corticosteroids
8. Histologic evidence of small cell carcinoma of the prostate.
9. Patients with a prior history of myocardial infarction, pulmonary embolism, CVA or atrial fibrillation.
10. Patients with active thrombophlebitis.
11. Patients with evidence of active angina as evidenced by chest pain responsive to sublingual nitroglycerin or other anginal equivalent.
12. Medical conditions, which, in the opinion of the investigators would jeopardize either the patient or the integrity of the data obtained
13. Patients who are currently receiving active therapy for other neoplastic disorders will not be eligible for study.
14. Patients taking any of the following medications who cannot discontinue these medications for three weeks during administration of androgen deprivation: aprepitant, bexarotene, clarithromycin, itraconazole, ketoconazole, St. John's wort.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is to evaluate the induction of tumor and prostate-specific immunity by androgen deprivation and estradiol administration. | End of Study

SECONDARY OUTCOMES:
Effects of androgen deprivation and estradiol administration on tumor infiltration by T lymphocytes, NK cells, and plasmacytoid dendritic cells | End of Study

CONTACTS AND LOCATIONS:
Overall Officials: R. Bruce Montgomery, MD, Principal Investigator — University of Washington; VA Puget Sound Health Care System
Locations (2):
- United States (2):
  - VA Puget Sound Health Care System, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington